CLINICAL TRIAL: NCT01506440
Title: Feasibility Study of a Cognitive Assessment Tool During Systemic Chemotherapy for Cancer Patients
Brief Title: Cognitive Assessments in Patients With Cancer Undergoing Chemotherapy
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00018421; NCI-2011-03034 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 99611 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2011-10-21; First posted 2012-01-10 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Malignant Neoplasm; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Neoplasms | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Supportive Care (cognitive assessment): Patients complete cognitive assessments, comprising HVLT-R, TMT-A, TMT-B, DSC, Animals, MoCA, and DST. Patients also complete the Beck Depression Inventory. Assessments are administered on day 1 of chemotherapy and at 6-8 weeks and 12-16 weeks after day 1 of chemotherapy.
  Interventions: Procedure: cognitive assessment; Procedure: quality-of-life assessment

INTERVENTIONS:
Procedure: cognitive assessment — Given cognitive assessments
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
This pilot clinical trial studies cognitive assessments in patients with cancer undergoing chemotherapy. Questionnaires that measure cognitive changes during chemotherapy may help identify the side effects of chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the feasibility of administering a cognitive assessment battery in a medical oncology clinic.

SECONDARY OBJECTIVES:

I. To estimate the variability of the various cognitive tests and to assess changes in cognitive performance based on the results of cognitive assessments obtained prior to chemotherapy and at 6 to 8 weeks and 12 to 16 weeks after the initiation of chemotherapy.

II. To explore the association of cognitive performance with the Eastern Cooperative Oncology Group (ECOG) performance status as evaluated by the patient's oncology team.

III. To assess the association between cognitive performance and the occurrence of a serious adverse event during chemotherapy.

OUTLINE:

Patients complete cognitive assessments, comprising Hopkins Verbal Learning Test-Revised (HVLT-R), Trail Making Test Parts A & B (TMT-A, TMT-B), Digit Symbol Coding Test (DSC), Category Fluency Test (Animals), Montreal Cognitive Assessment (MoCA), and Digit Span Test (DST). Patients also complete the Beck Depression Inventory. Assessments are administered on day 1 of chemotherapy and at 6-8 weeks and 12-16 weeks after day 1 of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed cancer
* Patients are candidates for systemic chemotherapy for their cancer diagnosis
* Life expectancy must be greater than 6 months
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had prior systemic chemotherapy in their lifetime
* Patients with known brain metastases should be excluded from this clinical trial because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* Patients may not be participating on any other study investigating cognitive function
* Patients who are non-English speaking are ineligible
* Patients with hematologic malignancies are ineligible
* Patients with primary central nervous system malignancies are ineligible

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being treated for the first time using standard chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Operational and logistical feasibility of administering cognitive assessment battery in medical oncology clinic environment during administration of chemotherapy. | Baseline to 16 weeks after the start of chemotherapy
  To determine whether cognitive assessment tools can be administered within the clinical and scheduling constraints of current chemotherapy administration practices.

SECONDARY OUTCOMES:
Changes in cognition over time | Baseline to 16 weeks after the start of chemotherapy
  As measured by cognitive assessment instruments
Association of cognitive performance with performance status and adverse events (AE) | Baseline to 16 weeks after the start of chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Klepin, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States